CLINICAL TRIAL: NCT04810559
Title: Near Patient Study of the OraQuick ADVANCE® HIV-1/2 Rapid Antibody Test in Oral Fluid and Fingerstick Whole Blood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REACH - HIV- OraQuick- 1.0
Record Dates: First submitted 2021-03-15; First posted 2021-03-23 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: HIV Testing; HIV Infections
Keywords: HIV; Testing; Point-of-care; OraQuick; Canada
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Cross-sectional, prospective, field trial (near patient study)
Masking Description: Subject enrollment is by unblinded staff and testing is by blinded healthcare providers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Investigational Device (Experimental)
  Interventions: Device: OraQuick ADVANCE® HIV-1/2 Rapid Antibody Test

INTERVENTIONS:
Device: OraQuick ADVANCE® HIV-1/2 Rapid Antibody Test — OraQuick ADVANCE® HIV-1/2 Rapid Antibody Test in oral fluid and fingerstick blood conducted by untrained healthcare providers compared to laboratory 4th generation Ag/Ab EIA results performed on venous blood.

SUMMARY:
Point-of-care (POC) tests for HIV are easy to use, rapid and provide accurate results while the patient is still in-front of a healthcare provider (HCP). Currently only blood-based POC tests for HIV are licensed for use in Canada. The OraQuick ADVANCE® HIV-1/2 Rapid Antibody Test is a POC test developed by OraSure Technologies, Inc. to detect HIV antibodies in oral fluid and fingerstick blood samples. As this device is very similar to the OraQuick HIV Self-Test, Health Canada requires evidence that HCPs can successfully perform the POC version of the OraQuick test in addition to performance of the self test version by intended users.

This study involves a minimum of 9 HCPs and 600 Patients at clinic sites in Toronto and Ottawa (Ontario), Montreal (Quebec) and Edmonton (Alberta). It will assess the OraQuick ADVANCE® Test's simplicity and accuracy in the hands of HCPs who have never used this Test.

To assess performance, using only the test kit instructions for use, HCPs will collect and test oral fluid and fingerstick blood samples from patients with the OraQuick ADVANCE® Test and will then read and interpret those results. Results of the OraQuick ADVANCE® Test will be compared with results of a venous blood sample collected from each patient and tested with a usual, licensed, laboratory test method.

To assess usability, HCPs will interpret various mock device test results and respond to a questionnaire to determine if the test instructions for use are clear and simple, that they are aware of test requirements and limitations and provide opinions on the ease of use of the test.

A final report of study results will be provided to the Test manufacturer for inclusion in the Health Canada license application process.

DETAILED DESCRIPTION:
Background and Rationale:

At the end of 2018, the Public Health Agency of Canada (PHAC) noted 2,242 new HIV infections (incidence rate of 6 per 100,000 people) representing a slight increase from 2016 estimates. For the same period, PHAC estimated there were 62,050 Canadians living with HIV (prevalence rate 167 per 100,000) and about 18,700 Canadians were missed throughout the HIV care continuum, including 8,300 who are living with HIV but were undiagnosed. This represents about 13% of Canadians living with HIV but are unaware of their status and not in care.

As testing is the entry point to HIV care, it is likely that those who are undiagnosed are not engaging in HIV testing services. PHAC's "Pan-Canadian Framework for Action " sets out an overarching and comprehensive approach to address sexually transmitted and blood-borne infections including HIV, and is composed of 26 opportunities for action, including enhancing testing. Testing opportunities which include elimination of barriers to access testing and normalization of testing through primary healthcare providers (HCPs), strategies that use community-based services and HIV self-testing could help Canada reach the undiagnosed. However, testing by HCPs within clinical settings remains the foundation to Canadian HIV care programs.

Point-of-care (POC) tests for HIV may have substantial utility for increased identification of HIV-infected individuals through their relative ease of use and portability, as well as their ability to deliver rapid, actionable results while the HCP still has access to the patient. OraSure Technologies, Inc. has developed a POC test, the OraQuick ADVANCE® HIV-1/2 Rapid Antibody Test, which requires no additional instrumentation and can be used by HCPs in multiple near patient settings. The OraQuick ADVANCE® Test is a single-use, visually read, qualitative, in vitro lateral flow immunoassay to detect antibodies to HIV-1 and HIV-2 in oral fluid and fingerstick blood. The Test package includes a specific step-by-step instructions, the device, testing buffer solution and a device stand. It is available in the United States (FDA approved) but is not currently approved for use in Canada.

Currently only blood-based POC tests for HIV are licensed for use in Canada. Having a licensed, oral-fluid test in addition to blood-based tests available for use in Canada provides another option to increase the uptake of HIV testing, and further increase the potential of reaching undiagnosed individuals living with HIV in Canada. Studies have shown that interest and acceptability of testing with oral fluid is high.

The objective of this near patient study is to demonstrate the simplicity and accuracy of the OraQuick ADVANCE® HIV-1/2 Rapid Antibody Test when used by untrained HCPs in a clinical setting. A secondary objective includes the ability of HCPs to correctly interpret a variety of contrived (mock) test device results.

Hypothesis: The OraQuickADVANCE® HIV-1/2 Rapid Antibody Test as performed by untrained HCPs will meet or exceed the accuracy, usability and label comprehension requirements from Health Canada for license as a Class IV in vitro diagnostic device for Canadian market entry.

Study Design:

This study was designed around the requirements set out in the Health Canada Guidance Document: "Guidance for Manufacturers of Human Immunodeficiency Virus (HIV) Rapid Diagnostic Tests (RDT's) for Use at Point of Care or Self Testing, 2017". It is a blinded, controlled study to evaluate the ability of HCPs to perform and interpret the results of the OraQuick ADVANCE® HIV-1/2 Rapid Antibody Test.

This protocol involves collection of oral fluid and fingerstick whole blood from approximately 600 patients to test with the OraQuick ADVANCE® Test device. Testing will be conducted by HCPs (blinded to patient's history and HIV diagnosis) in clinical settings. All patient participants will also have a venous blood sample collected (prior to fingerstick and oral fluid collection) for testing of plasma at a central laboratory with a 4th generation HIV Ag/Ab EIA (licensed for use in Canada) and positives will be confirmed using a standard HIV testing algorithm in place at the respective central laboratories. Results from the OraQuick ADVANCE® Test will be compared to results from the blood based 4th generation EIA. The sensitivity and specificity of the test result will be calculated relative to the confirmatory test process, where applicable. HCP qualification and assessment of the ease of device use will be evaluated. HCPs will also read and interpret 20 contrived (mock) device results in order to assess their ability to correctly interpret 5 potential test results, i.e. strong positive, weak positive, negative, invalid with no control and no test line, and invalid with no control and a positive test line.

Investigators will provide descriptive statistics for subject and HCP parameters. Test results will be compared to a Health Canada licensed 4th generation EIA test and investigators will calculate positive and negative percent agreement (with two-sided 95% confidence interval for both) for each matrix (fingerstick and oral fluid) separately. For mock device interpretation, agreement of the OraQuick ADVANCE® HIV-1/2 Rapid Antibody Test results with each sample type reactivity will be calculated overall and for each HCP operator. Safety will be assessed by the incidence of reported adverse events.

Sample population:

The study population requirements published by Health Canada for near patient studies of untrained HCP testers stipulates that the prospective study include: A minimum of 3 POC sites (different geographic locations), a minimum of 9 HCPs, 200 known HIV positive individuals and 400 individuals whose HIV status is unknown including 200 individuals at high risk of HIV infection (e.g. intravenous drug users, men who have sex with men, etc.). Self-reported practices or behaviour will be used to define those at high risk.

Hypothesis: The OraQuickADVANCE® HIV-1/2 Rapid Antibody Test as performed by untrained HCPs will meet or exceed the accuracy, usability and label comprehension requirements from Health Canada for license as a Class IV in vitro diagnostic device for Canadian market entry.

Study Design:

This study was designed around the requirements set out in the Health Canada Guidance Document: "Guidance for Manufacturers of Human Immunodeficiency Virus (HIV) Rapid Diagnostic Tests (RDT's) for Use at Point of Care or Self Testing, 2017". It is a blinded, controlled study to evaluate the ability of HCPs to perform and interpret the results of the OraQuick ADVANCE® HIV-1/2 Rapid Antibody Test.

This protocol involves collection of oral fluid and fingerstick whole blood from approximately 600 patients to test with the OraQuick ADVANCE® Test device. Testing will be conducted by HCPs (blinded to patient's history and HIV diagnosis) in clinical settings. All patient participants will also have a venous blood sample collected (prior to fingerstick and oral fluid collection) for testing of plasma at a central laboratory with a 4th generation HIV Ag/Ab EIA (licensed for use in Canada) and positives will be confirmed using a standard HIV testing algorithm in place at the respective central laboratories. Results from the OraQuick ADVANCE® Test will be compared to results from the blood based 4th generation EIA. The sensitivity and specificity of the test result will be calculated relative to the confirmatory test process, where applicable. HCP qualification and assessment of the ease of device use will be evaluated. HCPs will also read and interpret 20 contrived (mock) device results in order to assess their ability to correctly interpret 5 potential test results, i.e. strong positive, weak positive, negative, invalid with no control and no test line, and invalid with no control and a positive test line.

Investigators will provide descriptive statistics for subject and HCP parameters. Test results will be compared to a Health Canada licensed 4th generation EIA test and investigators will calculate positive and negative percent agreement (with two-sided 95% confidence interval for both) for each matrix (fingerstick and oral fluid) separately. For mock device interpretation, agreement of the OraQuick ADVANCE® HIV-1/2 Rapid Antibody Test results with each sample type reactivity will be calculated overall and for each HCP operator. Safety will be assessed by the incidence of reported adverse events.

Sample population:

The study population requirements published by Health Canada for near patient studies of untrained HCP testers stipulates that the prospective study include: A minimum of 3 POC sites (different geographic locations), a minimum of 9 HCPs, 200 known HIV positive individuals and 400 individuals whose HIV status is unknown including 200 individuals at high risk of HIV infection (e.g. intravenous drug users, men who have sex with men, etc.). Self-reported practices or behaviour will be used to define those at high risk.

Study Intervention Details:

HCPs will be recruited by site coordinators first. If HCPs are interested in participating they will complete the informed consent process and then complete an initial HCP questionnaire which will collect information such as demographics, occupation and POC device experience (about 15 minutes).

After this, patients will be recruited to the study when they come in for voluntary HIV testing (e.g. POC testing) and routine HIV follow-up care at study sites. If patients consent to participating, all those enrolled will voluntarily complete a questionnaire (collecting demographics and HIV medical history information) and then provide their venous whole blood sample (for clinical laboratory testing) and fingerstick and oral fluid specimens, for the testing with the OraQuick ADVANCE® Test - Visit 1 (day 1; about 40 - 60 minutes) as per protocol and study procedures. An unblinded HCP will administer the patient questionnaire and collect the venous whole blood sample. All patients will have a clinical laboratory test done for performance comparison using their venous sample, but only those with unknown HIV status will be instructed to return to the clinic for a follow-up visit two (2) weeks later to obtain their laboratory test results (Visit 2; about 10 - 15 minutes). Patients may also have a point-of-care (POC) test conducted on site as part of the clinic's standard of care testing, outside of the protocol and after all study procedures for Visit 1 are completed.

Two HCPs who are blinded to the patient history (including HIV diagnosis) will collect and test patient specimens, either the oral fluid or the fingerstick whole blood, using the OraQuick ADVANCE® Test by following the instructions provided in the Step-by-Step Instruction Guide and Package Insert for the Test. HCPs will then read, interpret (following the instruction guide) and document these test results for each patient. Sampling, testing and recording is estimated between 20 - 40 minutes per patient participant. At the end of testing at a site, HCPs will complete a second questionnaire which will include reading and interpreting 20 mock (contrived) device results, comprehension questions and collect information about ease of use and experience with the Test (about 1 hour).

ELIGIBILITY:
Healthcare provider Inclusion Criteria:

* Are at least 18 years of age
* Are able to provide informed consent
* Are paid employees of the study site(s)
* Are able to perform the study procedures outlined in the protocol

Healthcare provider Exclusion Criteria:

• Have used or watched someone use the OraQuick ADVANCE® HIV-1/2 Rapid Antibody Test

Patient Inclusion Criteria:

* Are at least 18 years of age
* Are able to provide informed consent
* Agree to provide accurate medical history
* Are able to provide up to 20mL blood by venipuncture, an oral fluid and a fingerstick blood sample
* Agree to undergo testing with the OraQuick ADVANCE® HIV-1/2 Rapid Antibody Test
* Patients with the known HIV positive status (diagnosis must be within five years of the study visit)
* Patients with unknown HIV status (last HIV negative test must be greater than 6 months prior to study visit)

Patient Exclusion Criteria:

* Are site employees
* Are in the judgment of the investigator unable to complete the study or are unlikely to comply with the study protocol; or
* Have been previously enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Percent Agreement | 1 year, year 1
  At the end of the study, positive and negative percent agreement (with two-sided 95% confidence interval for both) between OraQuick ADVANCE® HIV-1/2 Rapid Antibody Test and laboratory reference test for each matrix (fingerstick and oral fluid) will be calculated separately.
  For mock device interpretation, agreement of the OraQuick ADVANCE® HIV-1/2 Rapid Antibody Test results with each sample type reactivity will be calculated overall and for each healthcare provider test operator.

SECONDARY OUTCOMES:
Usability and Label comprehension | 1 year, year 1
  At the end of all testing, to assess usability, healthcare providers will interpret various mock device test results and respond to questionnaire to determine if the test instructions for use are clear and simple, that they are aware of test requirements and limitations and provide opinions on the ease of use of the test.

CONTACTS AND LOCATIONS:
Overall Officials: Sean B Rourke, PhD, Principal Investigator — MAP Centre for Urban Health Solutions, St. Micheal's Hospital
Locations (4):
- Canada (4):
  - Maple Leaf Research, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Women's Health in Women's Hands Community Health Centre, Toronto, Ontario
  - Clinique médicale l'Actuel, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No